CLINICAL TRIAL: NCT06640946
Title: Pain Control for Laser Epilation in Pilonidal Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: David Mooney (Other)
Responsible Party: Sponsor-Investigator, David Mooney, Associate Professor of Surgery, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P00048869
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Pilonidal Disease
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Placebo versus agent crossover per patient
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Cream will be applied by a clinician not involved in the laser procedure and will be removed prior to the procedure. Laser technicians will assess patient pain and will be blinded, as will the patient, to the study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Sham cream placed and then removed prior to laser follicle ablation.
  Interventions: Drug: Sham cream
- Active agent (Active Comparator): Topical lidocaine cream placed and then removed prior to laser follicle ablation.
  Interventions: Drug: Topical lidocaine

INTERVENTIONS:
Drug: Topical lidocaine — Topical lidocaine cream prior to laser follicle ablation
  Other Names: LMX
  Arms: Active agent
Drug: Sham cream — Placebo cream without lidocaine will be placed and removed before laser.
  Arms: Placebo

SUMMARY:
It's unclear if the application of topical lidocaine prior to laser follicle ablation is effective in reducing discomfort from the procedure. This study will use a doubly blinded case-control model to evaluate pain scores after the procedure comparing topical lidocaine to placebo.

DETAILED DESCRIPTION:
Patients presenting to a dedicated Pilonidal Care Clinic who have at least 2 future laser follicle ablations planned will be queried to determine their interest in participating in the study. Patients will be randomized to topical lidocaine or placebo, which will be applied for 30 minutes prior to the laser procedure, before which it will be removed. Laser technicians will be unaware of which cream the patient received and will record a post-procedure Likert pain score, from 0 to 10.

Patients will return in 6 to 8 weeks at which time they will crossover to the other group. Patients who received lidocaine cream will receive placebo and patients who received placebo will receive lidocaine cream. Cream removal and laser follicle ablation, with post-procedure pain score recording, will be conducted as during the first visit.

Twenty patients will be recruited and each patient will act as their own control.

ELIGIBILITY:
Inclusion Criteria: undergoing laser follicle ablation for pilonidal disease and expected to need at least 2 more treatments -

Exclusion Criteria: Unwilling to consent, not expected to need at least 2 more laser follicle ablations, not a candidate for laser

-

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Pain related to laser follicle ablation | 5 minutes
  Patient description on a Likert scale from 0 to 10 of the discomfort associated with the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley P Stoeckel, MD, Study Chair — Boston Children's
Locations (1):
- Boston Children's Hospital at Waltham, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Protocol details and anonymized patient data will be shared
Supporting Information: Study Protocol
Time Frame: 90 days after study completion, and for 1 year
Access Criteria: Investigator approval